CLINICAL TRIAL: NCT00908895
Title: Non-bridging Radio-radial Fixator Compared to Percutaneous Pinning for Unstable Distal Radius Fracture. A Prospective Randomized Trial.
Brief Title: Non-bridging Fixator Versus Percutaneous Pinning for Distal Radius Fractures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hopital de l'Enfant-Jesus (Other)
Responsible Party: Pelet Stéphane, MD, PhD, Hopital de l'Enfant-Jésus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEJ-206
Record Dates: First submitted 2009-05-26; First posted 2009-05-27 (Estimated); Results first posted 2010-06-07 (Estimated); Last update posted 2011-03-01 (Estimated); Status verified 2009-11

CONDITIONS: Radius Fractures
Keywords: Radius fractures; Radio-radial fixator; Percutaneous pinning; Grip strength
MeSH Terms: conditions — Radius Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radio-radial fixator (Experimental): Patients are operated on using a radio-radial fixator (Distal radius fixator, Synthes)
  Interventions: Procedure: Radio-radial fixator
- Percutaneous pinning (Active Comparator): Two K-wires inserted on a percutaneous way (dorsally and from the styloid), with a cast for 6 weeks
  Interventions: Procedure: Percutaneous pinning

INTERVENTIONS:
Procedure: Radio-radial fixator — Using the Distal Radius Fixator from Synthes. A single splint for 5 days.
  Arms: Radio-radial fixator
Procedure: Percutaneous pinning — Insert two K-wires in the distal radius, one in the fracture line dorsally and one from the styloid. A cast for 6 weeks.
  Arms: Percutaneous pinning

SUMMARY:
The treatment of extra-articular distal radius fractures is still controversial. In Canada, most patients with unstable fractures are treated with pinning and cast. Results are often associated with shortening and lack of function.

The purpose of the study is to compare stabilization with a radio-radial fixator to the usual method, suggesting that the radio-radial fixator will provide more strength at 6 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Distal radius fracture Frykman I or II
* Unstable fracture according to Lafontaine's criteria
* Fracture line more than 1cm form the joint line
* Closed fracture
* Age > 18 years
* Surgery performed between 72 hours from the trauma
* Monotrauma
* Patient signed the informed consent

Exclusion Criteria:

* Distal radius fracture Frykman III-VI (intra-articular fracture)
* Open fracture
* Polytraumatism
* Stable or non-displaced fracture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2003-04; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Département d'orthopédie, CHA-Pavillon Enfant-Jésus, Québec, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started in April of 2003 and finished in June of 2006.
Pre-assignment Details: Only surgical fractures were addressed to the research team, after prior selection by orthopedic surgeon. So we didn't see all radius fractures in the department.
Period: Overall Study
Arm/Group | Radio-radial Fixator | Percutaneous Pinning
Started | 57 | 63
Completed | 53 | 57
Not Completed | 4 | 6
Not completed — Lost to Follow-up | 1 | 3
Not completed — algodystrophy | 2 | 2
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Radio-radial Fixator | Percutaneous Pinning | Total
Number analyzed (Participants) | 57 | 63 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 51 | 97
  >=65 years | 11 | 12 | 23
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (19) | 54 (16) | 55.6 (18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 44 | 84
  Male | 17 | 19 | 36
Region of Enrollment [Number; unit: participants]
  Canada | 57 | 63 | 120

OUTCOME MEASURES:

1. Primary Outcome: The Grip Strength
Description: Grip strength measured with Jamar dynamometer in kilograms and adjusted to the opposite side in percentage. Correction made according to dominance.
Time Frame: 6 months
Population: No participant changed to the other group. Patients lost or with complications were not analyzed
Measure: Mean (95% Confidence Interval); unit: Percentage of opposite side
Arm/Group | Radio-radial Fixator | Percutaneous Pinning
Number analyzed (Participants) | 53 | 57
Percentage of opposite side | 98.3 [92.5 to 103.9] | 62.6 [56.1 to 68.9]
Statistical Analysis 1: Comparison: Radio-radial Fixator vs Percutaneous Pinning; We assess that 15% is a significative strength difference. According to a 80% study power, a SD at 25% and a 20% lost to follow-up, we found 118 patients for the all study; Test type: Superiority or Other; p < 0.05, Chi-squared; Cox Proportional Hazard = 70, Standard Deviation 25

2. Secondary Outcome: Range of Movement of Wrist
Description: Range of motion were divided in subgroups: dorsal flexion, volar flexion, pronation, supination, radial inclination, cubital inclination.
  Motion is described as a percentage of the opposite side.
Time Frame: 6 months
Measure: Mean (95% Confidence Interval); unit: Percentage of opposite side
Arm/Group | Radio-radial Fixator | Percutaneous Pinning
Number analyzed (Participants) | 53 | 57
Percentage of opposite side
  Dorsal flexion | 93.8 [90.7 to 96.9] | 81.7 [77.8 to 85.6]
  Volar flexion | 93.5 [90.4 to 96.6] | 74.7 [69.5 to 79.9]
  Pronation | 98 [96.7 to 99.3] | 90 [87.2 to 92.8]
  Supination | 90 [86.5 to 93.5] | 80 [75.9 to 84.1]
  Radial inclination | 90.7 [86.1 to 95.3] | 71.1 [64.9 to 77.3]
  Cubital inclination | 94 [89.1 to 98.9] | 65.6 [57.7 to 73.5]
Statistical Analysis 1: Comparison: Radio-radial Fixator vs Percutaneous Pinning; Test type: Superiority or Other; p < 0.05, Chi-squared; Cox Proportional Hazard = 90, 95% CI [80 to 100], Standard Deviation 10

ADVERSE EVENTS:
Arm/Group | Radio-radial Fixator | Percutaneous Pinning
Serious Adverse Events (participants affected / at risk) | 0/57 | 0/63
Other Adverse Events (participants affected / at risk) | 0/57 | 0/63

LIMITATIONS AND CAVEATS:
Very long time between the end of the study and the manuscript preparation due to temporarily lack of statistician and the need for some national associations that the study is not published before presentation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No